CLINICAL TRIAL: NCT00538083
Title: Dark Chocolate and Cocoa Ingestion and Endothelial Function: A Randomized, Placebo Controlled, Cross-over Trial
Brief Title: Cocoa and Endothelial Function in Adults With Elevated BMI
Acronym: Chocolate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); The Hershey Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2005-12
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cardioprotection
Keywords: Cocoa; Overweight adults; Endothelial function; Blood pressure; Cardiovascular disease risk; Dark chocolate; Sugar
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1, 2 (Experimental): acute phase, solid dark chocolate, placebo
  Interventions: Other: Chocolate
- 3, 4, 5 (Experimental): acute phase, sugared cocoa, sugar-free cocoa, placebo
  Interventions: Other: Chocolate
- 6, 7, 8 (Experimental): sustained phase, sugared cocoa, sugar-free cocoa, placebo
  Interventions: Other: Chocolate

INTERVENTIONS:
Other: Chocolate — 74 grams of single dose solid dark chocolate versus placebo
  Arms: 1, 2
Other: Chocolate — 22 grams of single dose sugared cocoa, sugar-free cocoa, and placebo
  Arms: 3, 4, 5
Other: Chocolate — 22 grams of sugared cocoa, sugar-free cocoa, & placebo given for six weeks
  Arms: 6, 7, 8

SUMMARY:
Cardiovascular disease is the leading cause of death in the United States. Studies have shown that obesity is an important risk factor for development of cardiovascular disease. Endothelial dysfunction, a pathologic feature of obesity, predicts the occurrence of cardiovascular disease. Recent research findings indicate that consumption of cocoa exerts cardioprotective effects, which include increasing HDL levels, reduction in systolic BP, inhibition of platelet aggregation/activity and activation of endothelial nitric oxide synthase.

Proposed is a randomized controlled trial consisting of 4 phases designed to examine the dose-response, and the acute and sustained effects of cocoa consumption on endothelial function as a marker of cardiovascular disease risk in 45 otherwise healthy adults with a BMI 25-35kg/m2.

DETAILED DESCRIPTION:
Endothelial function has been used extensively to evaluate the acute and chronic effects of foods and nutrients on cardiac risk and can provide a direct measurement of the effect of cocoa powder consumption on vascular physiology in healthy adults with BMI between 25-35 kg/m2.

To our knowledge, our study is the first to examine the dose response effects of sugar free, liquid, cocoa and solid, dark chocolate with sugar consumption on FMD, concentrating on individuals with elevated BMI. Given the current epidemic of obesity in the United States; its role as a risk factor in the development of cardiovascular disease; and the fact that cardiovascular disease is the leading cause of mortality in this country, examination of the cardio-protective effects of cocoa or dark chocolate in an at risk population is of considerable potential interest. Demonstrating that ingestion of cocoa may reverse damage caused to the endothelium may lead to new dietary recommendations that may help curb the prevalence of heart disease in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 30 -75
* BMI between 25-35 kg/m2
* waist circumference above 88 cms. in women and 102 cms. in men
* non-smoker
* no strenuous exercise at least 8 hours prior to scanning
* to facilitate recruitment individuals with diagnosed hypertension or hyperlipidemia will be included provided that they have been stable on their medications for three months, and can refrain from taking their medication 12 hours prior to BARS testing.

Exclusion Criteria:

* Failure to meet inclusion criteria
* anticipated inability to complete study protocol for any reason
* current eating disorder
* diagnosed coronary artery disease
* diabetes
* sleep apnea
* current or impending pregnancy
* insulin or glucose sensitizing medication use, vasoactive medication or nutriceutical use (glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators)
* regular use of high dose vitamin E or C and unable to discontinue for duration of the study
* regular use of fiber supplements and unable to discontinue for duration of the study
* restricted diets by choice (i.e. vegan, Atkins diet etc)
* allergy to cocoa or chocolate.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Endothelial Function(acute & sustained phase) | Single dose(acute phase), 6 weeks (sustained phase)

SECONDARY OUTCOMES:
Blood Pressure(acute and sustained phase), lipid profile(sustained), LDL oxidation(sustained), lipid hydroperoxide(sustained), CRP(sustained), blood glucose(sustained), body weight(sustained), waist circumference(sustained), endothelin(sustained) | Single dose(acute phase), 6 weeks(sustained phase)

CONTACTS AND LOCATIONS:
Overall Officials: David L Katz, MD, Principal Investigator — Yale-Griffin Prevention Research Center; Zubaida Faridi, MPH, Study Director — Yale-Griffin Prevention Research Center
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States